CLINICAL TRIAL: NCT02778477
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study To Assess The Safety, Tolerability And Pharmacokinetics Of Multiple Ascending Doses Of Pf-06423264 Administered Topically To Sequential Cohorts Of Healthy Subjects With And Without Oily Skin
Brief Title: Topical Multiple Ascending Dose Study for PF-06423264
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Preliminary analysis of accrued data failed to indicate any meaningful pharmacodynamic response.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Basic Science
Other Study IDs: B7561002; 2014-003736-39 (EudraCT Number)
Record Dates: First submitted 2016-05-17; First posted 2016-05-20 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Normal Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (18):
- Part A_Cohort 1_Active (Experimental): Multiple ascending dose of PF-06423264
  Interventions: Drug: PF-06423264
- Part A_Cohort 1_Placebo (Placebo Comparator): Multiple dose of placebo
  Interventions: Other: Placebo
- Part A_Cohort 2_Active (Experimental): Multiple ascending dose of PF-06423264
  Interventions: Drug: PF-06423264
- Part A_Cohort 2_Placebo (Placebo Comparator): Multiple dose of placebo
  Interventions: Other: Placebo
- Part A_Cohort 3_Active (Experimental): Multiple ascending dose of PF-06423264
  Interventions: Drug: PF-06423264
- Part A_Cohort 3_Placebo (Placebo Comparator): Multiple dose of placebo
  Interventions: Other: Placebo
- Part A_Cohort 4_Active (Experimental): Multiple ascending dose of PF-06423264
  Interventions: Drug: PF-06423264
- Part A_Cohort 4_Placebo (Placebo Comparator): Multiple dose of placebo
  Interventions: Other: Placebo
- Part A_Cohort 5_Active (Experimental): Multiple ascending dose of PF-06423264
  Interventions: Drug: PF-06423264
- Part A_Cohort 5_Placebo (Placebo Comparator): Multiple dose of placebo
  Interventions: Other: Placebo
- Part A_Cohort 6_Active (Experimental): Multiple ascending dose of PF-06423264
  Interventions: Drug: PF-06423264
- Part A_Cohort 6_Placebo (Placebo Comparator): Multiple dose of placebo
  Interventions: Other: Placebo
- Part A_Cohort 7_Active (Experimental): Multiple ascending dose of PF-06423264
  Interventions: Drug: PF-06423264
- Part A_Cohort 7_Placebo (Placebo Comparator): Multiple ascending dose of placebo
  Interventions: Other: Placebo
- Part B_Cohort 1_Active (Experimental): Multiple doses of PF-06423264
  Interventions: Drug: PF-06423264
- Part B_Cohort 1_Placebo (Placebo Comparator): Multiple doses of placebo
  Interventions: Other: Placebo
- Part B_Cohort 2_Active (Experimental): Multiple doses of PF-06423264
  Interventions: Drug: PF-06423264
- Part B_Cohort 2_Placebo (Placebo Comparator): Multiple doses of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-06423264 — Multiple ascending dose of PF-06423264
  Arms: Part A_Cohort 1_Active; Part A_Cohort 2_Active; Part A_Cohort 3_Active; Part A_Cohort 4_Active; Part A_Cohort 5_Active; Part A_Cohort 6_Active; Part A_Cohort 7_Active; Part B_Cohort 1_Active; Part B_Cohort 2_Active
Other: Placebo — Multiple dose of placebo
  Other Names: Placebo comparator
  Arms: Part A_Cohort 1_Placebo; Part A_Cohort 2_Placebo; Part A_Cohort 3_Placebo; Part A_Cohort 4_Placebo; Part A_Cohort 5_Placebo; Part A_Cohort 6_Placebo; Part A_Cohort 7_Placebo; Part B_Cohort 1_Placebo; Part B_Cohort 2_Placebo

SUMMARY:
The current study is the first clinical trial proposed with PF-06423264. It is designed to evaluate the safety, tolerability, and pharmacokinetics (PK) following administration of multiple ascending doses of PF-06423264 to healthy adult subjects with or without oily skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and female of non-childbearing potential;
* Body Mass Index 17.5-35.5 kg/m2;
* Body weight >50 kg;

Exclusion Criteria:

* Evidence of history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergises, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Number of Subjects With Treatment Emergent Treatment-Related Adverse Events (AEs) or other safety concerns | Baseline (Day 0) up to 28 days after last dose of study medication
  Assessment by adverse event monitoring, 12 lead ECGs, telemetry, vital signs and clinical safety laboratory measurements.
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a subject who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug was assessed by the investigator (Yes/No). Subjects with multiple occurrences of an AE within a category were counted once within the category.
Number of Participants with Draize-like scoring and clinical observation | Baseline (Day 1) up to Day 42+3
  Modified Draize-like scoring and clinical observation. Severity estimated by clinical signs and scoring; ranged 0-4: 0= No reaction visible, 1= Trace reaction - barely perceptible pinkness, 2= Mild reaction - readily visible pinkness, 3= Moderate reaction - definite redness, 4= Strong to severe reaction - very intense redness.
Number of Participants With Clinical Laboratory Abnormalities | Baseline (Day 0) up to 28 days after last dose
  Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, lactate dehydrogenase, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (sodium, potassium, chloride, calcium, phosphate, bicarbonate); clinical chemistry (glucose, creatine kinase); immunology (CRP); urinalysis (dipstick [urine specific gravity, decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, bilirubin], microscopy [urine RBC, WBC, urate crystals, calcium, oxalate, miscellaneous [urine mucus and leucocytes]).
Number of Participants With Abnormal Electrocardiogram (ECG) | Baseline (Day 0) up to 28 days after last dose
  Criteria for potential clinical concern in ECG parameters: Maximum QTcF interval (Fridericia's Correction) in range of 450 to less than 480 msec, maximum QTc interval increase from baseline in range of 30 to less than 60 msec and >=60 msec.
Number of Participants With Categorical Vital Signs Data | Baseline (Day 0) up to 28 days after last dose
  Number of participants with maximum increase from Baseline in sitting SBP and DBP of greater than or equal to 30 mmHg was reported.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for PF-06423264 | 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24 hours post dose on Day 1 and 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24, 36, and 48 hours post dose on Day 14
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Concentration for PF-06423264 | 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24 hours post dose on Day 1 and 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24, 36, and 48 hours post dose on Day 14
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for PF-06423264 | 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24 hours post dose on Day 1 and 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24, 36, and 48 hours post dose on Day 14
  Area under the concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 12 hours.
Plasma Decay Half-Life (t1/2) for PF-06423264 | 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24 hours post dose on Day 1 and 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24, 36, and 48 hours post dose on Day 14
  Plasma Decay Half-Life (t1/2)
Apparent Volume of Distribution (Vz/F) for PF-06423264 | 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24 hours post dose on Day 1 and 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24, 36, and 48 hours post dose on Day 14
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Apparent Total Body Clearance (CL/F) for | 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24 hours post dose on Day 1 and 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24, 36, and 48 hours post dose on Day 14
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after apparent total body clearance is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Observed Accumulation Ratio (Rac) for PF-06423264 | 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24 hours post dose on Day 1 and 0, 0.5, 1, 2, 4, 5, 6, 8, 12, 24, 36, and 48 hours post dose on Day 14
  Rac was calculated as, area under the curve from time zero to end of dosing interval on Day Y (AUCtau) divided by area under the curve from time zero to end of dosing interval on Day X(AUCtau).
change from baseline in sebum lipid components and sebum excretion | Baseline (Day 0) up to 16 days after last dose of study medication
  change from baseline in sebum lipid components and sebum excretion as assessed with Sebutape strips and Sebumeter measurements on the forehead of subjects with oily skin

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7561002&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Placebo-controlled+Study+To+Assess+The+Safety%2C+Tolerability+And+Pharmacokinetics+Of+Single+And++Multiple+Ascending+Doses+Of+Pf-06423264+Administered+Topically+To+Sequential+Cohorts+Of+Healthy+Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7561002&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Placebo-controlled+Study+To+Assess+The+Safety%2C+Tolerability+And+Pharmacokinetics+Of+Multiple+Ascending+Doses+Of+Pf-06423264+Administered+Topically+To+Sequential+Cohorts+Of+Healthy+Subjects+With+And+Without+Oily+Skin